CLINICAL TRIAL: NCT02772068
Title: Hemodynamic Response to Exercise in Heart Failure With Preserved Ejection Fraction (HFpEF) Patients After Upregulation of SERCA2a
Brief Title: Hemodynamic Response to Exercise in HFpEF Patients After Upregulation of SERCA2a
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Benjamin Levine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Benjamin Levine, Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STU 042013-039; R01AG017479 (NIH)
Record Dates: First submitted 2016-05-11; First posted 2016-05-13 (Estimated); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — Istaroxime; Exercise

STUDY DESIGN:
Intervention Model Description: Two separate groups of subjects (senior controls and patients with HFpEF) receiving istaroxime
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Senior Control (Active Comparator): Fifteen healthy senior subjects will perform light exercise at a fixed heart rate of 100 beats per minute. Subjects will then be given either placebo infusion (normal saline) or Istaroxime infusion for one hour. Subjects will be blinded to which infusion they are receiving. Subjects will then repeat light exercise at a fixed heart rate of 100 beats per minute. Primary outcome is changes in cardiac filling pressures during exercise.
  Interventions: Drug: Istaroxime; Other: Exercise
- Heart failure patients (Experimental): Fifteen HFpEF subjects will perform light exercise at a fixed heart rate of 100 beats per minute. Subjects will then be given either placebo infusion (normal saline) or Istaroxime infusion for one hour. Subjects will be blinded to which infusion they are receiving. Subjects will then repeat light exercise at a fixed heart rate of 100 beats per minute. Primary outcome is changes in cardiac filling pressures during exercise.
  Interventions: Drug: Istaroxime; Other: Exercise

INTERVENTIONS:
Drug: Istaroxime — Subjects will be given Istaroxime, a novel SERCA2a activator one hour prior and during exercise.
  Other Names: exercise
Other: Exercise

SUMMARY:
Heart failure with preserved ejection fraction or HFpEF, represents nearly 50% of all heart failure cases and is particularly common in the elderly. The disease has no current treatment options. Symptoms typically occur during exertion or exercise and is likely the result of increased cardiac and pulmonary congestion as a result of impaired diastolic function. Istaroxime is a novel activator of SERCA2a, an important regulator of calcium uptake within the myocyte. We will test the hypothesis that Istaroxime will improve diastolic function during exercise in HFpEF patients which in turn will reduce cardiac and pulmonary congestion.

DETAILED DESCRIPTION:
About half of all elderly patients with a diagnosis of congestive heart failure have apparently normal systolic function, so called "heart failure with a preserved ejection fraction" or HFpEF. To date, no effective therapy for HFpEF has been found, in part because of failure to discern key pathophysiologic pathways.

An extensive amount of pre-clinical work has identified that altered sarcoplasmic reticulum (SR) Ca2+ uptake, storage, and release play a major role in the changes in cardiac relaxation associated with aging, especially regarding sequestration of Ca++ by the sarcoplasmic reticular Ca++-ATPase (SERCA2a), which causes cardiac muscle relaxation by reducing cytosolic Ca++. Istaroxime is a relatively new drug that augments lusitropic function by upregulating SERCA2a activity in the heart.

Because of the clear importance of slowed relaxation in HFpEF, and the evidence that depressed SERCA2a activity contributes to the slowed relaxation with aging, the proposed study may be establish the "impairment of SERCA2a" hypothesis as a mechanism of impaired relaxation in HFpEF subjects.

ELIGIBILITY:
Healthy Senior Controls

Inclusion Criteria:

* age > 60 years

Exclusion Criteria:

* Coronary Ischemia
* No chronic medical problems
* BMI > 30 kg/m2

HFpEF Subjects

Inclusion Criteria:

* age > 60 years
* signs and symptoms of heart failure
* ejection fraction > 50%
* objective evidence of diastolic dysfunction

Exclusion Criteria:

* Coronary Ischemia
* Chronic Kidney Disease, stage 4 or greater
* Persistent atrial fibrillation
* Severe valvular disease
* BMI > 45 kg/m2

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change in cardiac filling pressures (pulmonary capillary wedge pressure) during exercise with Istaroxime | Immediate; 90 minutes after infusion
  Change in cardiac filling pressures (pulmonary capillary wedge pressure) during exercise with Istaroxime

SECONDARY OUTCOMES:
Change in cardiac relaxation time (isovolumic relaxation time) during exercise with Istaroxime | 90 minutes
  Change in cardiac relaxation time (isovolumic relaxation time) during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Levine, MD, Principal Investigator — UT Southwestern
Locations (1):
- The Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

REFERENCES:
- [Derived] Sarma S, MacNamara JP, Hieda M, Howden EJ, Lawley JS, Livingston S, Samels M, Levine BD. SERCA2a Agonist Effects on Cardiac Performance During Exercise in Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2023 Jul;11(7):760-771. doi: 10.1016/j.jchf.2023.02.006. Epub 2023 Apr 19. PMID 37086245